CLINICAL TRIAL: NCT01347814
Title: Does Domperidone, a D2-antagonist Alter Gastric Emptying Rates and Appetite Sensations in Healthy Adults?
Brief Title: Effect of 10mg Domperidone on Gastric Emptying of a High-fat Meal and Appetite Sensations in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Limerick (Other)
Collaborators: Irish Research Council (Other)
Responsible Party: Amir Shafat/Dr, University of Limerick
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: DompGastEmpt
Record Dates: First submitted 2011-05-03; First posted 2011-05-04 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2011-05

CONDITIONS: Diabetes Mellitus
Keywords: Domperidone; gastric emptying; obesity; diabetes mellitus; Domperidone/pharmacology; Pharmacologic Actions; Physiological Effects of Drugs; Gastrointestinal Agents; Humans
MeSH Terms: conditions — Diabetes Mellitus; Obesity | interventions — Domperidone; Homeopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Domperidone 10mg — 10mg domperidone tablet 30 minutes before a test-meal.
  Other Names: Motilium
Drug: Placebo — Homeopathic (Sugar) pill-Placebo
  Other Names: Homeopathic medicine; Silicea, 6c, Weleda, Derbyshire, UK

SUMMARY:
The purpose of this study is to determine whether domperidone was sufficient to accelerate gastric emptying of a high-fat solid meal and reduce satiety responses in a healthy adult population.

DETAILED DESCRIPTION:
This study aims to investigate the effect of domperidone on gastric emptying and appetite sensations in healthy subjects. Domperidone is a dopamine 2 (D2) receptor antagonist with claims of gastrointestinal tract pro-kinetic activity. Accelerated gastric emptying (GE) may lead to reduced satiation, increased food intake and is associated with obesity and diabetes mellitus. It is hypothesized that domperidone will increase gastric emptying rate and reduce satiety responses to a high-fat meal.

The effect of acute oral administration of 10 mg domperidone on gastric emptying of a high-fat pancake test meal, and subjective appetite sensations by visual analogue scale will be measured for six hours postprandially in a randomized, placebo-controlled, single-blinded manner in 13 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-40 years

Exclusion Criteria:

* History of gastrointestinal-related conditions, diabetes mellitus or cardiovascular disease

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2008-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Gastric emptying half time | 6.5 Hours post ingestion
  Determination of Gastric emptying of a high-fat test meal measured by octanoic acid breath test after acute administration of 10mg domperidone

SECONDARY OUTCOMES:
Appetite sensations | 6.5 hours post ingestion
  Determination of appetite sensations associated with ingestion of a high-fat test meal by visual analogue scale after acute administration of 10mg domperidone

CONTACTS AND LOCATIONS:
Overall Officials: Amir Shafat, Principal Investigator — University of Limerick
Locations (1):
- Department of Physical Education & Sport Sciences, University of Limerick, Limerick, Ireland

REFERENCES:
- [Background] Reddymasu SC, Soykan I, McCallum RW. Domperidone: review of pharmacology and clinical applications in gastroenterology. Am J Gastroenterol. 2007 Sep;102(9):2036-45. doi: 10.1111/j.1572-0241.2007.01255.x. Epub 2007 May 3. PMID 17488253
- [Derived] Markey O, Shafat A. Does domperidone, a D2-antagonist alter gastric emptying rates and appetite sensations in healthy adults with high-fat meal? A block-randomised, single-blind placebo-controlled study. Ir J Med Sci. 2012 Jun;181(2):215-9. doi: 10.1007/s11845-011-0785-2. Epub 2011 Nov 29. PMID 22124998